CLINICAL TRIAL: NCT06235567
Title: Comparison of Intracanalicular Steroid-eluting Insert (Dextenza) to Topical Steroid Eye Drops for the Postoperative Management of Corneal Collagen Crosslinking
Brief Title: Dextenza Versus Topical Steroid Eye Drops for Postoperative Management Following Corneal Crosslinking
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Maanasa Indaram, MD (Other)
Responsible Party: Sponsor-Investigator, Maanasa Indaram, MD, Associate Professor of Clinical Ophthalmology, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-40498
Record Dates: First submitted 2024-01-09; First posted 2024-02-01 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus | interventions — Calcium Dobesilate; prednisolone acetate; Ophthalmic Solutions

STUDY DESIGN:
Intervention Model Description: For group A, the study drug, DEXTNZA, is administered during the surgical procedure and the patient does not need to do any additional steps. For group B, the patient will administer the anti-inflammatory steroid drops on the same 4 week post-operative schedule that is commonly used in standard of care. They will do one drop of Pred Forte in the affected eye 4 times a day for a week, 3 times a day for the second week, 2 times a day for the third week, and once a day for the fourth week.
  The fellow eye will receive the alternate treatment when undergoing the procedure at a subsequent date at least 3 weeks following the first eye, and both within 45 days of the screening visit. Day 0 to Day 30 surgery and assessment schedule will be followed twice, once for each eye.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dextenza insert (Experimental): This is a prospective, open-label, single-center, randomized, investigator-sponsored clinical study to compare dexamethasone intracanalicular insert and corticosteroid drops for post-treatment in patients undergoing epithelium-off corneal collagen cross linking surgery. The participant's worse eye will be randomized to one of the two treatments, and the fellow eye will receive the alternate treatment when undergoing the procedure at a subsequent date at least three weeks later. There will be a baseline/screening visit, a surgical/ insertion visit for each eye, and follow up visits over 6 months, for a total of 10 visits per patient.
  The study drug, DEXTNZA, is administered during the surgical procedure and the patient does not need to do any additional steps.
  Interventions: Drug: Dextenza 0.4Mg Ophthalmic Insert
- topical prednisolone acetate 1% (PredForte) eye drops (Active Comparator): This is a prospective, open-label, single-center, randomized, investigator-sponsored clinical study to compare dexamethasone intracanalicular insert and corticosteroid drops for post-treatment in patients undergoing epithelium-off corneal collagen cross linking surgery. The participant's worse eye will be randomized to one of the two treatments, and the fellow eye will receive the alternate treatment when undergoing the procedure at a subsequent date at least three weeks later. There will be a baseline/screening visit, a surgical/ insertion visit for each eye, and follow up visits over 6 months, for a total of 10 visits per patient.
  The patient will administer the anti-inflammatory steroid drops on the same 4 week post-operative schedule that is commonly used in standard of care. They will do one drop of Pred Forte in the affected eye 4 times a day for a week, 3 times a day for the second week, 2 times a day for the third week, and once a day for the fourth week.
  Interventions: Drug: topical prednisolone acetate 1% (PredForte) eye drops

INTERVENTIONS:
Drug: Dextenza 0.4Mg Ophthalmic Insert — This insert allows for sustained release of dexamethasone onto the ocular surface over a period of 28 days. It requires a single application and eliminates the potential for noncompliance, difficulty in administration and poor accuracy. Dextenza has been FDA approved for post-operative pain and inflammation following ophthalmic surgery. The pivotal trials included patients undergoing cataract surgery, not CXL surgery. In addition, the age range did not include those of pediatric age.
  Arms: Dextenza insert
Drug: topical prednisolone acetate 1% (PredForte) eye drops — The patient will administer the anti-inflammatory steroid drops on the same 4 week post-operative schedule that is commonly used in standard of care. They will do one drop of Pred Forte in the affected eye 4 times a day for a week, 3 times a day for the second week, 2 times a day for the third week, and once a day for the fourth week.
  Arms: topical prednisolone acetate 1% (PredForte) eye drops

SUMMARY:
This study aims to compare the use of Dextenza, an FDA-approved intracanilular drug-eluting insert that is designed to deliver a tapered dose of dexamethasone to the ocular surface for 30 days, to the standard of care, or the use of a month-long topical prednisolone acetate 1% (PredForte) eye drops starting from four times daily. Following treatment, Dextenza resorbs and exits the nasolacrimal system without the need for removal. Three prior phase 3 clinical trials have demonstrated that Dextenza is equally efficacious to a month-long topical Pred Forte taper in the treatment of postoperative inflammation following cataract surgery. This proposed study strives to demonstrate the non-inferiority of using Dextenza to treat postoperative inflammation following corneal collagen crosslinking compared to standard of care eye drops in a randomized trial. By demonstrating Dextenza's non-inferiority to treatment postoperative inflammation, the investigators hope to provide an alternative modality of treatment to patients who are unable to cooperate with or tolerate postoperative topical eye drop regimens, allowing for improved adherence to necessary therapy and thus improved postoperative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* The study will enroll patients age 13 and up with progressive keratoconus (KCN) who are scheduled for bilateral epithelial off corneal collagen cross-linking (CXL) with Photrexa. A patient's study eye must meet the following criteria to be eligible for inclusion in the study:

  1. Progressive keratoconus as defined by increasing astigmatism and/or keratometry on corneal topography or tomography or increasing cylindrical error on refraction
  2. Patients requiring general anesthetic for the procedure
  3. Preoperative central corneal thickness of >= 400 microns

Exclusion Criteria:

* History of acute hydrops in treated eye
* History of pre-existing severe corneal scarring in the treated eye
* History of pre-existing glaucoma in the treated eye
* History of or pharmaceutical treatment of glaucoma or ocular hypertension and history or current spikes in intraocular pressure (IOP) in either eye.
* History of pre-existing ocular inflammation or infection (conjunctivitis, keratitis, uveitis, or retinitis) in treated eye
* Active infectious systemic disease
* Obstructed nasolacrimal duct in the study eye(s)
* Patients with a nasolacrimal duct smaller than 0.4 mm or greater than or equal to 1.0 mm.
* Patients with stenosis to the location where the insert will be placed should be excluded from the study, as the study team would not engage in surgical procedures to expand or surgically correct that region
* Hypersensitivity to dexamethasone
* Patients being treated with immunomodulating agents in the study eye(s)
* Patients being treated with immunosuppressants and/or oral steroids
* Patients with severe disease that warrants critical attention, deemed unsafe for the study by the investigator

Ages: 13 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Corneal haze | 1 months (30 days)
  Assess the efficacy of the dexamethasone insert compared to corticosteroid drops for post-treatment in patients who have had epithelium-off corneal collagen cross linking procedure.
  This will be assessed by
  -Postoperative corneal haze as measured by the Physician with a slit lamp biomicroscopy and graded on a scale of 0-4+ (0 = least haze ; 4= most haze)
Corneal re-epithelialization | 6 months (180 days)
  Assess the efficacy of the dexamethasone insert compared to corticosteroid drops for post-treatment in patients who have had epithelium-off corneal collagen cross linking procedure.
  This will be assessed by
  -Physician measured corneal re-epithelialization after bandage contact lens removal by slit lamp biomicroscopy.
Keratometry | 6 months (180 days)
  Assess the efficacy of the dexamethasone insert compared to corticosteroid drops for post-treatment in patients who have had epithelium-off corneal collagen cross linking procedure.
  This will be assessed by
  Postoperative keratometry values (diopters) as measured by corneal topography or Pentacam tomography. Comparing the pre- to post- operative values.
Infection | 6 months (180 days)
  Adverse event end point: Postoperative infection as measured at any visit.

SECONDARY OUTCOMES:
Comfort | 6 months (180 days)
  To determine the effect of dexamethasone intracanalicular insert through day 180 as measured by:
  - Patient comfort postoperatively as measured by a 0-10 scale and determined by asking the patient (0= no comfort; 10= maximum comfort)
Ocular Pain Assessment | 6 months (180 days)
  To determine the effect of dexamethasone intracanalicular insert through day 180 as measured by:
  - Patient pain postoperatively as measured by a 0-10 scale and determined by asking the patient (0= no pain ; 10= maximum pain)
Ease of insertion | 6 months (180 days)
  To determine the effect of dexamethasone intracanalicular insert through day 180 as measured by:
  - Physician ease of insertion as measured by a 0-5-point scale (0= easy insertion ; 5= difficult insertion)
Comparison of Ophthalmic Medications for Tolerability Questionnaire | 6 months (180 days)
  To determine the effect of dexamethasone intracanalicular insert through day 180 as measured by:
  - Patient's and caregivers' therapy of preference as measured by the Comparison of Ophthalmic Medications for Tolerability Questionnaire (COMTOL)
IOP spikes incidence | 6 months (180 days)
  To determine the effect of dexamethasone intracanalicular insert through day 180 as measured by:
  - Incidence of IOP spikes (IOP increased >or = 10mmHg from baseline) measured
Anterior segment OCT | 6 months (180 days)
  To determine the effect of dexamethasone intracanalicular insert through day 180 as measured by:
  - Anterior segment OCT findings mean change from baseline
Best Corrected Visual Acuity | 6 months (180 days)
  To determine the effect of dexamethasone intracanalicular insert through day 180 as measured by:
  - Best corrected visual acuity mean change from baseline as measured

CONTACTS AND LOCATIONS:
Overall Officials: Maanasa Indaram, MD, Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - Mission Bay Hospital, San Francisco, California
  - UCSF Pediatric Ophthalmology, San Francisco, California
  - Wayne and Gladys Center for Vision, San Francisco, California

IPD SHARING:
Plan to Share IPD: No